CLINICAL TRIAL: NCT04427501
Title: A Randomized, Double-blind, Placebo-Controlled, Phase 2/3 Study to Evaluate the Efficacy and Safety of LY3819253 and LY3832479 in Participants With Mild to Moderate COVID-19 Illness
Brief Title: A Study of LY3819253 (LY-CoV555) and LY3832479 (LY-CoV016) in Participants With Mild to Moderate COVID-19 Illness
Acronym: BLAZE-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AbCellera Biologics Inc. (Industry); Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 17947; J2W-MC-PYAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; etesevimab; bebtelovimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Some treatment arms are open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY3819253 (Experimental): 700 mg, 2800 mg, 7000 mg, LY3819253 administered intravenously (IV)
  Interventions: Drug: LY3819253
- LY3819253 + LY3832479 (Experimental): 350 mg, 700 mg, 2800 mg LY3819253 + 700 mg, 1400 mg, 2800 mg LY3832479 administered IV or subcutaneously (SQ)
  Interventions: Drug: LY3819253; Drug: LY3832479
- LY3819253 + LY3832479 (Pediatric Addendum, Arm 22) (Experimental): LY3819253 dose based upon weight (weight Group: ≥40 kilogram (kg) = 700 mg dose, >20 kg to <40 kg = 350 mg dose, >12 kg to 20 kg = 175 mg dose and 1.5 kg to 12 kg = 15 mg/kg dose) and LY3832479 dose based upon weight (weight Group: ≥40 kg = 1400 mg dose, >20 kg to <40 kg = 700 mg dose, >12 kg to 20 kg = 350 mg dose and 1.5 kg to 12 kg = 30 mg/kg dose) administered IV.
  Interventions: Drug: LY3819253; Drug: LY3832479
- LY3853113 (Pediatric Addendum, Arm 23) (Experimental): LY3853113 dose based upon weight (Weight Group: ≥3.3 to ≤12 kg = 3 mg/kg dose, >12 to ≤20 kg = 43.75 mg dose, >20 to <40 kg = 87.5 mg dose, ≥40 kg = 175 mg dose) administered IV.
  Interventions: Drug: LY3853113
- Placebo (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3819253 — Administered IV
  Other Names: LY-CoV555; Bamlanivimab
  Arms: LY3819253; LY3819253 + LY3832479; LY3819253 + LY3832479 (Pediatric Addendum, Arm 22)
Drug: LY3832479 — Administered IV
  Other Names: LY-CoV016; Etesevimab
  Arms: LY3819253 + LY3832479; LY3819253 + LY3832479 (Pediatric Addendum, Arm 22)
Drug: LY3853113 — Administered IV
  Other Names: bebtelovimab
  Arms: LY3853113 (Pediatric Addendum, Arm 23)
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure how well LY3819253 and LY3832479 work against the virus that causes COVID-19. LY3819253 and LY3832479 will be given to participants with early symptoms of COVID-19. Samples will be taken from the back of the nose to determine how much virus is in the body at various times during the study. Participation could last about 12 weeks and includes one required visit to the study site, with the remainder of assessments performed in the home or by phone.

Pediatric participants, with mild to moderate COVID-19 illness, will enroll in a single-arm (Arm 22), open-label addendum to evaluate the pharmacokinetics and safety of LY3819253 and LY3832479. Enrollment began on March 31, 2021, and completed on September 24, 2021.

Pediatric participants, with mild to moderate COVID-19 illness, will enroll in a single-arm (Arm 23), open-label addendum to evaluate the pharmacokinetics and safety of LY3853113. Enrollment began on August 19, 2022, and completed on February 21, 2023.

ELIGIBILITY:
Inclusion Criteria:

* Are currently not hospitalized. (Not applicable to participants in treatment arm 22.)
* Have one or more mild or moderate COVID-19 symptoms: Fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, or shortness of breath with exertion. (Not applicable to participants in treatment arm 22.)
* Must have sample taken for test confirming viral infection no more than 3 days prior to starting the drug infusion
* Are males or females, including pregnant females who agree to contraceptive requirements
* Understand and agree to comply with planned study procedures
* Agree to the collection of nasopharyngeal swabs and venous blood. (Not applicable to participants in treatment arms 20-21.)
* The participant or legally authorized representative give signed informed consent and/or assent

Participants in treatment arms 7-9, 13-14, and 18-21 ONLY

* Are greater than or equal to (≥)18 years of age and must satisfy at least one of the following at the time of screening

  * Are pregnant
  * Are ≥65 years of age
  * Have a body mass index (BMI) ≥35
  * Have chronic kidney disease (CKD)
  * Have type 1 or type 2 diabetes
  * Have immunosuppressive disease
  * Are currently receiving immunosuppressive treatment or
  * Are ≥55 years of age AND have:

    * cardiovascular disease (CVD), OR
    * hypertension, OR
    * chronic obstructive pulmonary disease (COPD) or other chronic respiratory disease
* Are 12-17 years of age (inclusive) AND satisfy at least one of the following at the time of screening

  * Are pregnant
  * Have a body mass index (BMI) ≥85th percentile for their age and gender based on CDC growth charts, https://www.cdc.gov/growthcharts/clinical_charts.htm
  * Have sickle cell disease
  * Have congenital or acquired heart disease
  * Have neurodevelopmental disorders, for example, cerebral palsy
  * Have a medical-related technological dependence, for example, tracheostomy, gastrostomy, or positive pressure ventilation (not related to COVID-19)
  * Have asthma or reactive airway or other chronic respiratory disease that requires daily medication for control
  * Have type 1 or type 2 diabetes
  * Have chronic kidney disease
  * Have immunosuppressive disease, or
  * Are currently receiving immunosuppressive treatment

Participants in treatment arm 22 ONLY

- Are 0 (≥ 32 weeks gestational age AND ≥ 1.5 kilograms [kg]) to 17 years of age (inclusive) AND satisfy at least one of the following risk factors at the time of screening

* Are pregnant
* Have a BMI ≥85th percentile for their age and gender based on CDC growth charts, https://www.cdc.gov/growthcharts/clinical_charts.htm
* Have sickle cell disease
* Have congenital or acquired heart disease
* Have neurodevelopmental disorders, for example, cerebral palsy, autism, or Down syndrome (FAIR Health 2020; Spreat et al. 2020)
* Have a medical-related technological dependence, for example, tracheostomy, gastrostomy, or positive pressure ventilation (not related to COVID-19)
* Have asthma, cystic fibrosis, reactive airways disease or other chronic respiratory disease that requires daily medication for control
* Have type 1 or type 2 diabetes
* Have chronic kidney disease
* Have immunosuppressive disease, or
* Are currently receiving immunosuppressive treatment, or
* Are less than (<) one year of age.
* Have one or more COVID-19 symptoms

  * Shortness of breath/difficulty breathing
  * Fever
  * Sore throat
  * Nausea
  * Diarrhea
  * Tiredness
  * Headache
  * New loss of taste
  * Nasal congestion/runny nose
  * Chills
  * Stomachache
  * Vomiting
  * Cough
  * Muscle/body aches and pain
  * New loss of smell
  * Poor appetite or poor feeding (in babies)

Participants in treatment arm 23 ONLY:

Must have first positive result sample of current SARS-CoV-2 viral infection ≤3 days prior to start of treatment administration.

Participant can have COVID previously and still meet criteria for this addendum. Positive result needs to be from a current infection.

Are 0 (≥ 38 weeks gestational age and ≥ 3.3 kg) to <12 years of age at the time of screening, or are 12 to 17 and weighing <40 kg; and

* Have mild to moderate COVID-19 disease, including one or more COVID-19 symptoms within the last 7 days
* Shortness of breath/difficulty breathing
* Fever
* Sore throat
* Nausea
* Diarrhea
* Tiredness
* Headache
* New loss of taste
* Nasal congestion/runny nose
* Chills
* Malaise
* Vomiting
* Cough
* Muscle/body aches and pain
* New loss of smell
* Poor appetite or poor feeding (in babies under 1 year old)

Exclusion Criteria:

* Have oxygen saturation (SpO2) less than or equal to (≤)93 percent (%) on room air at sea level or ratio of arterial oxygen partial pressure (PaO2 in millimeters of mercury) to fractional inspired oxygen (FiO2) less than (<)300, respiratory rate greater than or equal to (≥)30 per minute, heart rate ≥125 per minute due to COVID-19
* Require mechanical ventilation or anticipated impending need for mechanical ventilation due to COVID-19
* Have known allergies to any of the components used in the formulation of the interventions
* Have hemodynamic instability requiring use of pressors within 24 hours of randomization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
* Have any co-morbidity requiring surgery within <7 days, or that is considered life-threatening within 29 days
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study
* Have a history of a positive SARS-CoV-2 test prior to the one serving as eligibility for this study
* Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing
* Have received treatment with a SARS-CoV-2 specific monoclonal antibody
* Have received convalescent COVID-19 plasma treatment
* Have participated in a previous SARS-CoV-2 vaccine study or have received a SARS-CoV-2 vaccine
* Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed
* Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Mothers who are breast feeding

Participants in Treatment Arm 22 ONLY

* Have a diagnosis of Multisystem Inflammatory Syndrome in Children (MIS-C) in the opinion of the investigator
* Are currently hospitalized for treatment of COVID-19. Other reasons for hospitalization are acceptable.

Participants in treatment arm 23 ONLY

* SpO2 ≤ 93% on room air at sea level, or while on chronic oxygen therapy and/or respiratory support due to underlying non-COVID-19 related comorbidity, respiratory rate ≥30 per minute, and heart rate ≥125 per minute due to COVID-19 (FDA February 2021)
* Require mechanical ventilation or anticipated impending need for mechanical ventilation due to COVID-19
* Have known allergies to any of the components used in the formulation of the interventions
* Have hemodynamic instability requiring use of pressors within 24 hours of randomization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
* Have any co-morbidity requiring surgery within 7 days, or that is considered life-threatening within 29 days
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study.
* Have received treatment with a SARS-CoV-2 specific monoclonal antibody or remdesivir within 90 days before dosing.
* Have received convalescent COVID-19 plasma treatment within 90 days before dosing
* Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed
* Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are currently pregnant or breast feeding

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3307 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - Clinnova Research - Redondo Beach, Redondo Beach, California
  - Bio-Medical Research, LLC, Miami, Florida
  - Rophe Adult and Pediatric Medicine, Union City, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - U of MA Mem Med Ctr, Worcester, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Sky Clinical Prime and Health Wellness Clinic, Fayette, Mississippi
  - Sky Clin Resch - Quinn HC, Ridgeland, Mississippi
  - Monroe Biomed Research, Monroe, North Carolina
  - B S & W Med Center, Dallas, Texas
  - Sun Research Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
URL: http://vivli.org/

REFERENCES:
- [Derived] Patel DR, Macpherson L, Bohm M, Upadhyaya H, Deveau C, Nirula A, Klekotka P, Williams M, Hufford MM. Efficacy and Safety of Low-Dose, Rapidly Infused Bamlanivimab and Etesevimab: Phase 3 BLAZE-1 Trial for Mild-to-Moderate COVID-19. Infect Dis Ther. 2024 Oct;13(10):2123-2134. doi: 10.1007/s40121-024-01031-z. Epub 2024 Sep 4. PMID 39230829
- [Derived] Upadhyaya HP, Chien JY, Long AJ, Bohm MS, Kallewaard NL, Macpherson LF, Patel DR, Hufford MM, Krull CJ, Ang JY, Chen P, Muller WJ, Potts JA, Quinn T, Williams M; BLAZE-1 Investigators. Pharmacokinetics, Efficacy, and Safety of a SARS-CoV-2 Antibody Treatment in Pediatric Participants: An Open-Label Addendum of a Placebo-Controlled, Randomized Phase 2/3 Trial. Infect Dis Ther. 2023 Jul;12(7):1861-1873. doi: 10.1007/s40121-023-00832-y. Epub 2023 Jun 17. PMID 37329415
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Chen P, Behre G, Hebert C, Kumar P, Farmer Macpherson L, Graham-Clarke PL, De La Torre I, Nichols RM, Hufford MM, Patel DR, Naegeli AN. Bamlanivimab and Etesevimab Improve Symptoms and Associated Outcomes in Ambulatory Patients at Increased Risk for Severe Coronavirus Disease 2019: Results From the Placebo-Controlled Double-Blind Phase 3 BLAZE-1 Trial. Open Forum Infect Dis. 2022 Apr 7;9(5):ofac172. doi: 10.1093/ofid/ofac172. eCollection 2022 May. PMID 35493124
- [Derived] Dougan M, Azizad M, Mocherla B, Gottlieb RL, Chen P, Hebert C, Perry R, Boscia J, Heller B, Morris J, Crystal C, Igbinadolor A, Huhn G, Cardona J, Shawa I, Kumar P, Blomkalns A, Adams AC, Van Naarden J, Custer KL, Knorr J, Oakley G, Schade AE, Holzer TR, Ebert PJ, Higgs RE, Sabo J, Patel DR, Dabora MC, Williams M, Klekotka P, Shen L, Skovronsky DM, Nirula A. A Randomized, Placebo-Controlled Clinical Trial of Bamlanivimab and Etesevimab Together in High-Risk Ambulatory Patients With COVID-19 and Validation of the Prognostic Value of Persistently High Viral Load. Clin Infect Dis. 2022 Aug 24;75(1):e440-e449. doi: 10.1093/cid/ciab912. PMID 34718468
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Nathan R, Shawa I, De La Torre I, Pustizzi JM, Haustrup N, Patel DR, Huhn G. A Narrative Review of the Clinical Practicalities of Bamlanivimab and Etesevimab Antibody Therapies for SARS-CoV-2. Infect Dis Ther. 2021 Dec;10(4):1933-1947. doi: 10.1007/s40121-021-00515-6. Epub 2021 Aug 10. PMID 34374951
- [Derived] Meng X, Wang P, Xiong Y, Wu Y, Lin X, Lu S, Li R, Zhao B, Liu J, Zeng S, Zeng L, Wu Y, Lu Y, Zhang J, Liu D, Wang S, Lu H. Safety, tolerability, pharmacokinetic characteristics, and immunogenicity of MW33: a Phase 1 clinical study of the SARS-CoV-2 RBD-targeting monoclonal antibody. Emerg Microbes Infect. 2021 Dec;10(1):1638-1648. doi: 10.1080/22221751.2021.1960900. PMID 34346827
- [Derived] Dougan M, Nirula A, Azizad M, Mocherla B, Gottlieb RL, Chen P, Hebert C, Perry R, Boscia J, Heller B, Morris J, Crystal C, Igbinadolor A, Huhn G, Cardona J, Shawa I, Kumar P, Adams AC, Van Naarden J, Custer KL, Durante M, Oakley G, Schade AE, Holzer TR, Ebert PJ, Higgs RE, Kallewaard NL, Sabo J, Patel DR, Dabora MC, Klekotka P, Shen L, Skovronsky DM; BLAZE-1 Investigators. Bamlanivimab plus Etesevimab in Mild or Moderate Covid-19. N Engl J Med. 2021 Oct 7;385(15):1382-1392. doi: 10.1056/NEJMoa2102685. Epub 2021 Jul 14. PMID 34260849
- [Derived] Gottlieb RL, Nirula A, Chen P, Boscia J, Heller B, Morris J, Huhn G, Cardona J, Mocherla B, Stosor V, Shawa I, Kumar P, Adams AC, Van Naarden J, Custer KL, Durante M, Oakley G, Schade AE, Holzer TR, Ebert PJ, Higgs RE, Kallewaard NL, Sabo J, Patel DR, Klekotka P, Shen L, Skovronsky DM. Effect of Bamlanivimab as Monotherapy or in Combination With Etesevimab on Viral Load in Patients With Mild to Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2021 Feb 16;325(7):632-644. doi: 10.1001/jama.2021.0202. PMID 33475701
- [Derived] Chen P, Nirula A, Heller B, Gottlieb RL, Boscia J, Morris J, Huhn G, Cardona J, Mocherla B, Stosor V, Shawa I, Adams AC, Van Naarden J, Custer KL, Shen L, Durante M, Oakley G, Schade AE, Sabo J, Patel DR, Klekotka P, Skovronsky DM; BLAZE-1 Investigators. SARS-CoV-2 Neutralizing Antibody LY-CoV555 in Outpatients with Covid-19. N Engl J Med. 2021 Jan 21;384(3):229-237. doi: 10.1056/NEJMoa2029849. Epub 2020 Oct 28. PMID 33113295
- See also: A Study of LY3819253 (LY-CoV555) and LY3832479 (LY-CoV016) in Participants With Mild to Moderate COVID-19 Illness (BLAZE-1) — https://trials.lillytrialguide.com/en-US/trial/63aASRmBPQCBCOfy5oO0er

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study has three parts: Phase 2, Phase 3 and pediatrics addendum. All participants in Placebo for Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab are also in Placebo For Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab therefore the two arms are combined to avoid double counting.
Groups:
- Phase 2: Placebo; Phase 3: Placebo; Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab: Participants received Placebo administered intravenously (IV).
- Phase 2: 700 mg Bamlanivimab: Participants received 700 milligram (mg) bamlanivimab administered IV.
- Phase 2: 2800 mg Bamlanivimab: Participants received 2800 mg bamlanivimab administered IV.
- Phase 2: 7000 mg Bamlanivimab: Participants received 7000 mg bamlanivimab administered IV.
- Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab: Participants received 2800 mg bamlanivimab and 2800 mg etesevimab administered IV.
- Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab: Participants received 700 mg bamlanivimab and 1400 mg etesevimab administered IV.
- Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab: Participants received 350 mg bamlanivimab and 700 mg etesevimab administered IV.
- Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22): Pediatric participants received a Bamlanivimab + Etesevimab dose based upon weight (Bamlanivimab dose: weight Group: ≥40 kg = 700 mg dose, >20 kg to <40 kg = 350 mg dose, >12 kg to 20 kg = 175 mg dose and 1.5 kg to 12 kg = 15 mg/kg dose) and Etesevimab dose: weight Group: ≥40 kg = 1400 mg dose, >20 kg to <40 kg = 700 mg dose, >12 kg to 20 kg = 350 mg dose and 1.5 kg to 12 kg = 30 mg/kg dose) administered IV.
- Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23): Pediatric participants received Bebtelovimab dose based upon weight (Weight Group: ≥3.3 to ≤12 kg = 3 mg/kg dose, >12 to ≤20 kg = 43.75 mg dose, >20 to <40 kg = 87.5 mg dose, ≥40 kg = 175 mg dose) administered IV.
Period: Overall Study
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23)
Started | 156 | 101 | 107 | 101 | 112 | 776 (Participants in Placebo for Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab and Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab were combined to avoid double counting.) | 518 | 513 | 141 | 213 | 94 | 17
Received at Least One Dose of Study Drug | 156 | 101 | 107 | 101 | 112 | 776 | 518 | 513 | 141 | 213 | 94 | 17
Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | 0 | 0 | 0 | 0 | 0 | 517 | 0 | 0 | 0 | 0 | 0 | 0
Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | 0 | 0 | 0 | 0 | 0 | 776 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 141 | 95 | 103 | 98 | 103 | 719 | 485 | 496 | 135 | 207 | 88 | 16
Not Completed | 15 | 6 | 4 | 3 | 9 | 57 | 33 | 17 | 6 | 6 | 6 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 5 | 1 | 2 | 0 | 2 | 11 | 10 | 10 | 2 | 5 | 2 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 2 | 2 | 3 | 7 | 25 | 15 | 7 | 4 | 1 | 4 | 0
Not completed — Other - as reported by the investigator | 1 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Phase 2: 700 mg Bamlanivimab: Participants received 700 mg bamlanivimab administered IV.
- Total: Total of all reporting groups
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23) | Total
Number analyzed (Participants) | 156 | 101 | 107 | 101 | 112 | 776 | 518 | 513 | 141 | 213 | 94 | 17 | 2849
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (15.38) | 43.5 (16.21) | 44.4 (14.61) | 45.7 (16.28) | 43.9 (16.39) | 53.4 (16.52) | 54.3 (17.08) | 54.5 (16.77) | 53.6 (15.70) | 52.7 (17.49) | 9.9 (4.76) | 26.19 (15.95) | 51.9 (16.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 63 | 51 | 58 | 58 | 404 | 279 | 265 | 68 | 108 | 43 | 9 | 1491
  Male | 71 | 38 | 56 | 43 | 54 | 372 | 239 | 248 | 73 | 105 | 51 | 8 | 1358
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 49 | 47 | 39 | 42 | 226 | 149 | 139 | 36 | 53 | 13 | 4 | 866
  Not Hispanic or Latino | 87 | 52 | 60 | 62 | 70 | 548 | 368 | 373 | 104 | 160 | 80 | 13 | 1977
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 3 | 0 | 0 | 15
  Asian | 8 | 1 | 5 | 3 | 2 | 33 | 16 | 18 | 6 | 6 | 0 | 0 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 6
  Black or African American | 7 | 7 | 7 | 8 | 4 | 61 | 44 | 41 | 16 | 28 | 67 | 12 | 302
  White | 133 | 90 | 90 | 89 | 105 | 667 | 449 | 445 | 116 | 175 | 22 | 5 | 2386
  More than one race | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 3 | 0 | 12
  Unknown or Not Reported | 5 | 0 | 3 | 1 | 1 | 7 | 6 | 3 | 1 | 1 | 2 | 0 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 156 | 101 | 107 | 101 | 112 | 776 | 518 | 513 | 141 | 213 | 94 | 17 | 2849
SARS-CoV-2 Viral Load [Mean (Standard Deviation); unit: Cycle threshold (Ct)] — Population: All participants who received at least one dose of study drug and had at least 1 post-baseline viral load measurement. Cycle threshold (Ct) denotes how many PCR cycles are required before the SARS-CoV-2 viral RNA reached a detectable level. Higher Ct values correspond to a lower viral load.
  Cycle threshold (Ct)
    number analyzed (Participants) | 152 | 101 | 107 | 101 | 109 | 774 | 508 | 510 | 141 | 213 | 86 | 16 | 2818
    (all) | 23.79 (7.78) | 23.80 (6.55) | 24.47 (7.61) | 23.42 (6.78) | 22.72 (8.01) | 24.26 (8.194) | 23.98 (8.22) | 24.15 (7.28) | 24.29 (6.82) | 25.62 (7.33) | 26.61 (7.458) | 28.79 (7.053) | 24.16 (7.75)

OUTCOME MEASURES:

1. Primary Outcome: Phase 3: Percentage of Participants Who Experience COVID-Related Hospitalization or Death From Any Cause in 2800 mg Bamlanivumab/2800 mg Etesevimab, 700 mg Bamlanivimab/1400mg Etesevimab and Their Placebo Groups
Description: COVID-19 Related Deterioration (yes/no) was defined as a participant experiencing COVID-19-related hospitalization (defined as 24 hours of acute care) or death from any cause by Day 29.
Time Frame: Baseline through Day 29
Population: Phase 3: All randomized participants who received at least one dose of study drug and had COVID-related hospitalization or death from any cause data available in arms Placebo, 2800 mg Bamlanivimab + 2800 mg Etesevimab and 700 mg Bamlanivimab + 1400 mg Etesevimab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab; Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab: Participants received Placebo administered intravenously (IV).
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab
Number analyzed (Participants) | 517 | 518 | 776 | 511
percentage of participants | 7.0 [4.8 to 9.2] | 2.1 [0.9 to 3.4] | 6.8 [5.1 to 8.6] | 0.8 [0.0 to 1.5]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.15 to 0.58]
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.12, 95% CI 2-sided [0.04 to 0.31]

2. Primary Outcome: Phase 3: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than a Prespecified Threshold in Arms 350 mg Bamlanivimab/700 mg Etesevimab and Placebo
Description: SARS-CoV-2 persistent high viral load (yes/no) was defined as ribonuclease P(RP) normalized viral load >=5.27 vs otherwise.
Time Frame: Day 7
Population: Phase 3: All randomized participants who received at least one dose of study drug and had non-missing viral load values in arms Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab and 350 mg Bamlanivimab + 700 mg Etesevimab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 141 | 213
percentage of participants | 34.8 [26.9 to 42.6] | 10.8 [6.6 to 15.0]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.13 to 0.40]

3. Primary Outcome: Phase 2: Change From Baseline to Day 11 in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load
Description: SARS-CoV-2 viral load was based on nasopharyngeal swab sampling for reverse transcription polymerase chain reaction (RT-PCR) testing for SARS-CoV-2. Least squares (LS) mean values were determined using a mixed-effects model repeated-measures (MMRM) that included log base 10 transformed baseline as a covariate, treatment, day, treatment-by-day interaction as fixed effects. If Day 11 SARS-CoV-2 viral load was missing, the earliest measurement closest to the Day 11 visit, but within 4 days (Day 7-Day 15), was used for the Day 11 value. If no measurements were available, the Day 11 viral load was treated as missing at random (MAR) in the analysis.
  Viral load is reported as normalized viral load and is unitless.
Time Frame: Baseline, Day 11
Population: Phase 2: All randomized participants who received at least one dose of study drug and had a baseline and day 11 viral load value.
Measure: Least Squares Mean (Standard Error); unit: unitless
Groups:
- Part A: Placebo: Participants received Placebo administered intravenously (IV).
Arm/Group | Part A: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 146 | 100 | 103 | 95 | 102
unitless | -3.80 (0.141) | -3.72 (0.170) | -4.08 (0.168) | -3.49 (0.175) | -4.37 (0.169)
Statistical Analysis 1: Comparison: Part A: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.6921, Mixed Models Analysis; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.35 to 0.52], Standard Error of Mean 0.221
Statistical Analysis 2: Comparison: Part A: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.2110, Mixed Models Analysis; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.71 to 0.16], Standard Error of Mean 0.219
Statistical Analysis 3: Comparison: Part A: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.1630, Mixed Models Analysis; Mean Difference (Net) = 0.31, 95% CI 2-sided [-0.13 to 0.76], Standard Error of Mean 0.225
Statistical Analysis 4: Comparison: Part A: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.0099, Mixed Models Analysis; Mean Difference (Net) = -0.57, 95% CI 2-sided [-1.00 to -0.14], Standard Error of Mean 0.220

4. Primary Outcome: Phase 2: Percentage of Participants Who Experience a Serious Adverse Event(s) SAE(s)
Description: An SAE was defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other different situations will have medical or scientific judgment to determine if they are SAE. A summary of SAEs and other non-serious adverse events (AEs), regardless of causality are reported in the Adverse Events section.
Time Frame: Baseline through Day 85
Population: Phase 2: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 156 | 101 | 107 | 101 | 112
percentage of participants | 0.6 | 0 | 0 | 0 | 0.9

5. Primary Outcome: Phase 3 and Phase 2/3 [Arm 22], Pharmacokinetics (PK): Mean Concentrations of LY3819253 (Bamlanivimab)
Description: Mean Concentration of Bamlanivimab in the presence of Etesevimab is reported. Due to the limited number of pediatric participants across all study arms in phase 3, PK concentration summary data was combined including phase 3 and phase 2/3 (Pediatric addendum, Arm 22) reporting arms. All pediatric participants from Phase 3 trial arms including Arm 22 who contributed data to the required outcome (PK concentration at Day 29) were included in the PK summary.
Time Frame: Day 29 Post-dose
Population: Phase 2/3: All randomized participants who received a complete dose of Bamlanivimab and Etesevimab and had an evaluable PK sample on Day 29.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- Phase 3 and Phase 2/3 (Pediatric Addendum, Arm 22): Bamlanivimab + Etesevimab: Pediatric participants from Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab reporting arms and Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) received a single weight category-dependent dose of the combination Bamlanivimab + Etesevimab dose based upon weight (Bamlanivimab dose: weight Group: ≥40 kg = 700 mg dose, >20 kg to <40 kg = 350 mg dose, >12 kg to 20 kg = 175 mg dose and 1.5 kg to 12 kg = 15 mg/kg dose) and Etesevimab dose: weight Group: ≥40 kg = 1400 mg dose, >20 kg to <40 kg = 700 mg dose, >12 kg to 20 kg = 350 mg dose and 1.5 kg to 12 kg = 30 mg/kg dose) administered IV.
Arm/Group | Phase 3 and Phase 2/3 (Pediatric Addendum, Arm 22): Bamlanivimab + Etesevimab
Number analyzed (Participants) | 95
micrograms per milliliter (μg/mL)
  Bamlanivimab 700 mg: Weight Group: ≥40 kg: number analyzed (Participants) | 64
  Bamlanivimab 700 mg: Weight Group: ≥40 kg | 29.9 (54.4)
  Bamlanivimab 350 mg: Weight Group: >20 kg to <40 kg: number analyzed (Participants) | 18
  Bamlanivimab 350 mg: Weight Group: >20 kg to <40 kg | 23.7 (45.6)
  Bamlanivimab 175 mg: Weight Group: >12 kg to 20 kg: number analyzed (Participants) | 10
  Bamlanivimab 175 mg: Weight Group: >12 kg to 20 kg | 21.2 (74.0)
  Bamlanivimab 15 mg/kg: Weight Group: 1.5 kg to 12 kg: number analyzed (Participants) | 3
  Bamlanivimab 15 mg/kg: Weight Group: 1.5 kg to 12 kg | 40.2 (23.2)

6. Primary Outcome: Phase 3 and Phase 2/3 [Arm 22], Pharmacokinetics (PK): Mean Concentrations of LY3832479 (Etesevimab)
Description: Mean Concentration of Etesevimab in the presence of Bamlanivimab is reported. Due to the limited number of pediatric participants across all study arms in phase 3, PK concentration summary data was combined including phase 3 and phase 2/3 (Pediatric addendum, Arm 22) reporting arms. All pediatric participants from Phase 3 trial arms including Arm 22 who contributed data to the required outcome (PK concentration at Day 29) were included in the PK summary.
Time Frame: Day 29 Post-dose
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Phase 3 and Phase 2/3 (Pediatric Addendum, Arm 22): Bamlanivimab + Etesevimab
Number analyzed (Participants) | 96
micrograms per milliliter (μg/mL)
  Etesevimab 1400 mg: Weight Group: ≥40 kg: number analyzed (Participants) | 65
  Etesevimab 1400 mg: Weight Group: ≥40 kg | 140 (44.0)
  Etesevimab 700 mg: Weight Group: >20 kg to <40 kg: number analyzed (Participants) | 18
  Etesevimab 700 mg: Weight Group: >20 kg to <40 kg | 129 (36.7)
  Etesevimab 350 mg: Weight Group: >12 kg to 20 kg: number analyzed (Participants) | 10
  Etesevimab 350 mg: Weight Group: >12 kg to 20 kg | 122 (57.3)
  Etesevimab 30 mg/kg: Weight Group: 1.5 kg to 12 kg: number analyzed (Participants) | 3
  Etesevimab 30 mg/kg: Weight Group: 1.5 kg to 12 kg | 193 (11.0)

7. Primary Outcome: Phase 2/3, PK: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) for Bebtelovimab [Arm 23]
Description: AUC0-∞ for Bebtelovimab was reported.
Time Frame: Day 60 Post-dose
Population: Phase 2/3: All randomized participants who received a complete dose of Bebtelovimab and had at least 1 post-dose PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23)
Number analyzed (Participants) | 16
microgram*day per milliliter (μg*day/mL) | 481 (45.8)

8. Secondary Outcome: Phase 3: Percentage of Participants Demonstrating Symptom Resolution
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and changes in taste and smell. Each symptom was scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Symptom resolution (yes/no) is defined as a score of 0 for shortness of breath, feeling feverish, body aches and pains, sore throat, chills, and headache; and a score of 0 or 1 for cough and fatigue on the symptom questionnaire (excluding the loss of appetite and changes in taste and smell symptoms). Missing data were imputed using non-responder imputation (NRI) method.
Time Frame: Day 11
Population: Phase 3: All randomized participants who received at least one dose of study drug and had non-missing Symptom Resolution values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 499 | 508 | 774 | 510 | 141 | 213
percentage of participants | 52.1 [47.7 to 56.5] | 61.2 [57.0 to 65.5] | 50.9 [47.4 to 54.4] | 61.8 [57.5 to 66.0] | 51.8 [43.5 to 60.0] | 63.8 [57.4 to 70.3]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.13 to 1.86]
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.24 to 1.95]
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.06 to 2.53]

9. Secondary Outcome: Phase 3: Percentage of Participants Demonstrating Symptom Improvement
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and changes in taste and smell. Each symptom will be scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Symptom improvement was defined as a participant experiencing both: Symptoms on the symptom questionnaire scored as moderate or severe at baseline are subsequently scored as mild or absent, and symptoms on the symptom questionnaire scored as mild or absent at baseline are subsequently scored as absent. Missing data were imputed using NRI method.
Time Frame: Day 11
Population: Phase 3: All randomized participants who received at least one dose of study drug and had non-missing Symptom Improvement values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 499 | 508 | 774 | 510 | 141 | 213
percentage of participants | 40.9 [36.6 to 45.2] | 51.0 [46.6 to 55.3] | 40.1 [36.6 to 43.5] | 52.7 [48.4 to 57.1] | 38.3 [30.3 to 46.3] | 54.0 [47.3 to 60.7]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.17 to 1.93]
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.33 to 2.09]
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.22 to 2.9]

10. Secondary Outcome: Phase 3: Percentage of Participants Who Experience COVID-Related Hospitalization, COVID-Related Emergency Room (ER) Visit, or Death From Any Cause
Description: COVID-19 Related Deterioration (yes/no) is defined as a patient experiencing COVID-19-related hospitalization, Emergency Room Visit, or Death from any causes vs otherwise.
Time Frame: Baseline through Day 85
Population: Phase 3: All randomized participants who received at least one dose of study drug and had COVID-related hospitalization, COVID-Related Emergency Room (ER) Visit, or death from any cause data available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 517 | 518 | 716 | 511 | 141 | 231
percentage of participants | 7.2 [4.9 to 9.4] | 2.5 [1.2 to 3.9] | 7.0 [5.2 to 8.7] | 1.2 [0.2 to 2.1] | 4.3 [0.9 to 7.6] | 0.9 [0.0 to 2.2]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.18 to 0.64]
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.07 to 0.38]
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.06 to 1.05]

11. Secondary Outcome: Phase 3: Change From Baseline to Day 7 in SARS-CoV-2 Viral Load
Description: Change from baseline to Day 7 (±2 days) in SARS-CoV-2 viral load was based on nasopharyngeal swab sampling for reverse transcription polymerase chain reaction (RT-PCR) testing for SARS-CoV-2. Least squares (LS) mean values were determined using a mixed-effects model repeated-measures (MMRM) that included log base 10 transformed baseline as a covariate, treatment, day, treatment-by-day interaction as fixed effects. If Day 7 SARS-CoV-2 viral load was missing, the earliest measurement closest to the Day 7 visit, but within 2 days (Day 5-Day 9), was used for the Day 7 value. If no measurements are available, the Day 7 viral load was treated as missing at random (MAR) in the analysis.
  Viral load is reported as normalized viral and is unitless.
Time Frame: Baseline, Day 7
Population: Phase 3: All randomized participants who received at least one dose of study drug and had a baseline and day 7 viral load value.
Measure: Least Squares Mean (Standard Error); unit: unitless
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 403 | 455 | 614 | 399 | 122 | 194
unitless | -2.46 (0.095) | -3.66 (0.090) | -2.56 (0.079) | -3.65 (0.098) | -2.51 (0.185) | -3.50 (0.147)
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p < 0.0000000, Mixed Models Analysis; Mean Difference (Net) = -1.20, 95% CI 2-sided [-1.46 to -0.94]
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; p < 0.0000000, Mixed Models Analysis; Mean Difference (Net) = -1.09, 95% CI 2-sided [-1.34 to -0.85]
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; p = 0.00003777, Mixed Models Analysis; Mean Difference (Net) = -0.99, 95% CI 2-sided [-1.45 to -0.52]

12. Secondary Outcome: Phase 3: Time to Sustained Symptom Resolution
Description: Sustained symptom resolution was defined as 2 consecutive assessments with a score of 0 for shortness of breath, feeling feverish, body aches and pains, sore throat, chills, and headache; and a score of 0 or 1 for cough and fatigue on the symptom questionnaire. Participants who did not experience sustained symptom resolution by completion or early discontinuation of study were censored at the date of their last visit during. Additionally, participants who were hospitalized were censored at their date of hospitalization.
Time Frame: Baseline through Day 29
Population: Phase 3: All randomized participants (including censored) who received at least one dose of study drug and who had at least one post-baseline symptom measurement. Participants censored: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab = 121, 2800 mg Bamlanivimab + 2800 mg Etesevimab = 88, Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab= 226, 700 mg Bamlanivimab + 1400 mg Etesevimab= 128, Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab=44, 350 mg Bamlanivimab + 700 mg Etesevimab=43
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 499 | 508 | 774 | 510 | 141 | 213
Days | 9.00 [8.00 to 10.00] | 8.00 [7.00 to 8.00] | 9.00 [9.00 to 10.00] | 8.00 [7.00 to 9.00] | 9.00 [8.00 to 13.00] | 6.00 [5.00 to 8.00]
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.007, Stratified Log-rank; Hazard Ratio (HR) = 1.213
Statistical Analysis 2: Comparison: Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab vs Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab; Test type: Superiority; p = 0.130, Stratified Log-rank; Hazard Ratio (HR) = 1.111
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; p = 0.012, Stratified Log-rank; Hazard Ratio (HR) = 1.380

13. Secondary Outcome: Phase 3: Time to SARS-CoV-2 Viral Clearance
Description: Participants who did not experience SARS-CoV-2 viral clearance by completion or early discontinuation of study were censored at the date of their last visit.
Time Frame: Baseline through Day 29
Population: Phase 3: All randomized participants (Including censored) who received at least 1 dose of study drug and had at least 1 post-baseline viral load measurement. Censored participants: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab = 358, 2800 mg Bamlanivimab + 2800 mg Etesevimab = 325, Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab =530, 700 mg Bamlanivimab + 1400 mg Etesevimab= 326, Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab=95, 350 mg Bamlanivimab + 700 mg Etesevimab=114
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo For 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab
Number analyzed (Participants) | 499 | 508 | 774 | 510 | 141 | 213
Days | NA [NA to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe. | NA [NA to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe. | NA [NA to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe. | NA [NA to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe. | NA [NA to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe. | NA [14.00 to NA] — Median cannot be calculated due to insufficient number of events occurring within the timeframe.
Statistical Analysis 1: Comparison: Phase 3: Placebo For 2800 mg Bamlanivimab + 2800 mg Etesevimab vs Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.007, Stratified Log-rank; Hazard Ratio (HR) = 1.355
Statistical Analysis 2: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; p = 0.033, Stratified Log-rank; Hazard Ratio (HR) = 1.237
Statistical Analysis 3: Comparison: Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab vs Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab; Test type: Superiority; p = 0.017, Stratified Log-rank; Hazard Ratio (HR) = 1.521

14. Secondary Outcome: Phase 2: Change From Baseline to Day 11 in SARS-CoV-2 Viral Load Among Participants Enrolled With Recent Symptoms Prior to Randomization
Description: SARS-CoV-2 viral load was based on nasopharyngeal swab sampling for reverse transcription polymerase chain reaction (RT-PCR) testing for SARS-CoV-2. This analysis included only participants whose symptoms developed no more than 8 days prior to randomization. Least squares (LS) mean values were determined using a mixed-effects model repeated-measures (MMRM) that included log base 10 transformed baseline as a covariate, treatment, day, treatment-by-day interaction as fixed effects. If Day 11 SARS-CoV-2 viral load is missing, the earliest measurement closest to the Day 11 visit, but within 4 days (Day 7-Day 15), will be used for the Day 11 value. If no measurements are available, the Day 11 viral load will be treated as MAR in the analysis.
Time Frame: Baseline, Day 11
Population: Phase 2: All randomized participants who received at least one dose of study drug and had baseline and post-baseline viral load value. Participants enrolled with recent symptoms prior to randomization.
Measure: Least Squares Mean (Standard Error); unit: unitless
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 123 | 84 | 88 | 81 | 95
unitless | -4.03 (0.155) | -3.87 (0.187) | -4.20 (0.184) | -3.65 (0.191) | -4.46 (0.178)
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.499, Mixed Models Analysis; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.31 to 0.64], Standard Error of Mean 0.243
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.492, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.64 to 0.31], Standard Error of Mean 0.241
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.125, Mixed Models Analysis; Mean Difference (Net) = 0.38, 95% CI 2-sided [-0.11 to 0.86], Standard Error of Mean 0.246
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.069, Mixed Models Analysis; Mean Difference (Net) = -0.43, 95% CI 2-sided [-0.89 to 0.03], Standard Error of Mean 0.236

15. Secondary Outcome: Phase 2: Percentage of Participants Demonstrating Symptom Resolution
Description: Symptoms associated with COVID-19 were evaluated using a questionnaire that contains the following symptoms: cough, shortness of breath, feeling feverish, fatigue, body aches and pain, sore throat, chills, headache, loss of appetite, and changes in taste and smell. Each symptom will be scored daily by the participant as experienced during the past 24 hours with following rating and score: None or absent (0), Mild (1), Moderate (2) and Severe (3). Symptom resolution was defined as all symptoms (those scored 0-3) on the symptom questionnaire scored as absent (0). Symptom Resolution (yes/no) was defined as all symptoms (excluding the loss of appetite and changes in taste and smell symptoms) on the symptom questionnaire scored as absent vs otherwise.
  Missing data were imputed using non-responder imputation (NRI) method.
Time Frame: Day 11
Population: Phase 2: All randomized participants who received at least one dose of study drug and had non-missing Symptom Resolution values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 152 | 101 | 107 | 101 | 109
percentage of participants | 36.8 [29.2 to 44.5] | 50.5 [40.7 to 60.2] | 40.2 [30.9 to 49.5] | 43.6 [33.9 to 53.2] | 45.9 [36.5 to 55.2]
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.034, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.04 to 2.90]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.594, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.69 to 1.91]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.291, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.79 to 2.20]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.143, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.88 to 2.40]

16. Secondary Outcome: Phase 2: Percentage of Participants Demonstrating Symptom Improvement
Description: as for outcome 9
Time Frame: Day 11
Population: Phase 2: All randomized participants who received at least one dose of study drug and had non-missing Symptom Improvement values
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 152 | 101 | 107 | 101 | 109
percentage of participants | 43.4 [35.5 to 51.3] | 59.4 [49.8 to 69.0] | 44.9 [35.4 to 54.3] | 58.4 [48.8 to 68.0] | 53.2 [43.8 to 62.6]
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.014, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.14 to 3.15]
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.828, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.64 to 1.74]
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.022, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.09 to 3.02]
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.119, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.90 to 2.43]

17. Secondary Outcome: Phase 2, Pharmacokinetics (PK): Mean Concentration of Bamlanivimab Alone and in the Presence of Etesevimab
Description: (PK): Mean Concentration of Bamlanivimab alone and in the Presence of Etesevimab
Time Frame: Day 29 Post-dose
Population: Phase 2: All randomized participants who received a complete dose of Bamlanivimab (for Bamlanivimab only arms) or Bamlanivimab in the Presence of Etesevimab (for Bamlanivimab + Etesevimab) and had at least 1 post-dose PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter (µg/mL)
Groups:
- Phase 2: 700 mg Bamlanivimab: Participants received 700 mg bamlanivimab (alone) administered IV.
- Phase 2: 2800 mg Bamlanivimab: Participants received 2800 mg bamlanivimab (alone) administered IV.
- Phase 2: 7000 mg Bamlanivimab: Participants received 7000 mg bamlanivimab (alone) administered IV..
Arm/Group | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 80 | 89 | 86 | 92
Microgram/milliliter (µg/mL) | 25.6 (42.2) | 83.8 (50.0) | 227 (39.6) | 100 (46.1)

18. Secondary Outcome: Phase 2, PK: Mean Concentration of Etesevimab in the Presence of Bamlanivimab
Description: PK: Mean Concentration of Etesevimab in the Presence of Bamlanivimab
Time Frame: Day 29 Post-dose
Population: Phase 2: All randomized participants who received a complete dose of Etesevimab in the Presence of Bamlanivimab and had at least 1 post-dose PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 92
µg/mL | 243 (35.1)

19. Secondary Outcome: Phase 2: Percentage of Participants Who Experience COVID-Related Hospitalization, COVID-Related Emergency Room (ER) Visit, or Death From Any Cause
Description: Percentage of Participants Who Experience COVID-Related Hospitalization, COVID-Related ER Visit, or Death from Any Cause
Time Frame: Baseline through Day 85
Population: Phase 2: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 156 | 101 | 107 | 101 | 112
percentage of participants | 5.8 [2.1 to 9.4] | 1.0 [0.0 to 2.9] | 1.9 [0.0 to 4.4] | 2.0 [0.0 to 4.7] | 0.9 [0.0 to 2.6]
Statistical Analysis 1: Comparison: Part A: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.098, Regression, Logistic; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.04 to 1.31]
Statistical Analysis 2: Comparison: Part A: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.165, Regression, Logistic; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.09 to 1.51]
Statistical Analysis 3: Comparison: Part A: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.191, Regression, Logistic; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.10 to 1.60]
Statistical Analysis 4: Comparison: Part A: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.075, Regression, Logistic; Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.04 to 1.18]

20. Secondary Outcome: Phase 2: Time to SARS-CoV-2 Viral Clearance
Description: as for outcome 13
Time Frame: Baseline through Day 29
Population: Phase 2: All randomized participants (including censored) who received at least one dose of study drug and had at least one post-baseline viral load measurement. Censored: Part A: Placebo= 68, Phase 2: 700 mg Bamlanivimab=39, Phase 2: 2800 mg Bamlanivimab=40, Phase 2: 7000 mg Bamlanivimab=42 and Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab=45
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab
Number analyzed (Participants) | 152 | 101 | 107 | 101 | 109
Days | 24 [22.00 to NA] — Some upper bound confidence intervals were not estimable due to insufficient events occurring within the timeframe. | 25.00 [21.00 to 27.00] | 23.00 [19.00 to 25.00] | 25.00 [22.00 to NA] — Some upper bound confidence intervals were not estimable due to insufficient events occurring within the timeframe. | 21.00 [17.00 to NA] — Some upper bound confidence intervals were not estimable due to insufficient events occurring within the timeframe.
Statistical Analysis 1: Comparison: Phase 2: Placebo vs Phase 2: 700 mg Bamlanivimab; Test type: Superiority; p = 0.616, Stratified Log-rank
Statistical Analysis 2: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab; Test type: Superiority; p = 0.281, Stratified Log-rank
Statistical Analysis 3: Comparison: Phase 2: Placebo vs Phase 2: 7000 mg Bamlanivimab; Test type: Superiority; p = 0.815, Stratified Log-rank
Statistical Analysis 4: Comparison: Phase 2: Placebo vs Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab; Test type: Superiority; p = 0.334, Stratified Log-rank

21. Secondary Outcome: Phase 2/3: Percentage of Participants Who Experience COVID-19 Related Hospitalization, COVID-Related Emergency Room (ER) Visit, or Death From Any Cause [Arm 22]
Description: as for outcome 19
Time Frame: Baseline through Day 29
Population: Phase 2/3: All randomized participants who received at least one dose of study drug and had COVID-related hospitalization, COVID-Related Emergency Room (ER) Visit, or death from any cause data available.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 94
percentage of participants | 0

22. Secondary Outcome: Phase 2/3: Change From Baseline to Day 7 in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load [Arm 22]
Description: SARS-CoV-2 viral load was based on nasopharyngeal swab sampling for reverse transcription polymerase chain reaction (RT-PCR) testing for SARS-CoV-2.
  Viral load is reported as normalized viral load and is unitless.
Time Frame: Baseline, Day 7
Population: Phase 2/3: All randomized participants who received at least one dose of study drug and had a baseline and day 7 viral load value.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 84
unitless | -4.37 (2.740)

23. Secondary Outcome: Phase 2/3: Percentage of Participants With SARS-CoV-2 Viral Load Greater Than a Prespecified Threshold [Arm 22]
Description: SARS-CoV-2 persistent high viral load (yes/no) is defined as RP normalized viral load >5.27 vs otherwise. Percentage of response is calculated by n/Nx*100% (n = number of participants in the specified category, Nx = number of participants with non-missing values)
Time Frame: Day 7
Population: Phase 2/3: All randomized participants who received at least one dose of study drug and had a day 7 viral load value.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 92
percentage of participants | 10.9

24. Secondary Outcome: Phase 2/3: Time to Complete Symptom Resolution [Arm 22]
Description: Complete symptom resolution was defined as absence of all symptoms at a single timepoint.
Time Frame: Baseline through Day 29
Population: Phase 2/3: All randomized participants (including censored) who received at least one dose of study drug and had non-missing Symptom Resolution values. Censored participants = 7.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 94
days | 5.00 [4.00 to 6.00]

25. Secondary Outcome: Phase 2/3: Time to Sustained Complete Symptom Resolution [Arm 22]
Description: Sustained complete symptom resolution is defined as the first of 2 consecutive days with complete symptom resolution.
Time Frame: Baseline through Day 29
Population: Phase 2/3: All randomized participants (including censored) who received at least one dose of study drug and had non-missing Symptom Resolution values. Censored participants = 13.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 94
days | 7.00 [5.00 to 8.00]

26. Secondary Outcome: Phase 2/3: Time to SARS-CoV-2 Viral Clearance [Arm 22]
Description: as for outcome 13
Time Frame: Baseline through Day 29
Population: Phase 2/3: All randomized participants (Including censored) who received at least one dose of study drug and had at least one post-baseline viral load measurement. Censored participants = 34.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22)
Number analyzed (Participants) | 94
days | 11.00 [8.00 to 13.00]

ADVERSE EVENTS:
Time Frame: Baseline Up to 85 Days
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly. Phase2/3 Pediatric Arms did not collect adverse events by dose.
Groups:
- Phase 3: Placebo; Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab: Participants received Placebo administered IV.
Arm/Group | Phase 2: Placebo | Phase 2: 700 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab | Phase 2: 7000 mg Bamlanivimab | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab | Phase 3: Placebo | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23)
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/101 | 0/107 | 0/101 | 0/112 | 0/518 | 15/776 | 0/513 | 0/141 | 0/213 | 0/94 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/156 | 2/101 | 0/107 | 0/101 | 1/112 | 10/518 | 8/776 | 16/513 | 4/141 | 1/213 | 1/94 | 0/17
Other Adverse Events (participants affected / at risk) | 44/156 | 29/101 | 26/107 | 24/101 | 23/112 | 72/518 | 92/776 | 61/513 | 17/141 | 14/213 | 16/94 | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 2: Placebo (N=156) | Phase 2: 700 mg Bamlanivimab (N=101) | Phase 2: 2800 mg Bamlanivimab (N=107) | Phase 2: 7000 mg Bamlanivimab (N=101) | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab (N=112) | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab (N=518) | Phase 3: Placebo (N=776) | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab (N=513) | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab (N=141) | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab (N=213) | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) (N=94) | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23) (N=17)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 1/279 (1) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Uterine mass (Reproductive system and breast disorders) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 1/404 (1) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 2: Placebo (N=156) | Phase 2: 700 mg Bamlanivimab (N=101) | Phase 2: 2800 mg Bamlanivimab (N=107) | Phase 2: 7000 mg Bamlanivimab (N=101) | Phase 2: 2800 mg Bamlanivimab + 2800 mg Etesevimab (N=112) | Phase 3: 2800 mg Bamlanivimab + 2800 mg Etesevimab (N=518) | Phase 3: Placebo (N=776) | Phase 3: 700 mg Bamlanivimab + 1400 mg Etesevimab (N=513) | Phase 3: Placebo For 350 mg Bamlanivimab + 700 mg Etesevimab (N=141) | Phase 3: 350 mg Bamlanivimab + 700 mg Etesevimab (N=213) | Phase 2/3: Bamlanivimab + Etesevimab (Pediatric Addendum, Arm 22) (N=94) | Phase 2/3: Bebtelovimab (Pediatric Addendum, Arm 23) (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye paraesthesia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xanthopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 3 (3) | 4 (4) | 4 (4) | 4 (5) | 5 (5) | 5 (5) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0/71 (0) | 0/38 (0) | 0/56 (0) | 0/43 (0) | 0/54 (0) | 0/239 (0) | 1/372 (1) | 0/248 (0) | 0/73 (0) | 0/105 (0) | 0/51 (0) | 0/8 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1/85 (1) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 1/279 (1) | 1/404 (1) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 1/68 (1) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/85 (0) | 0/63 (0) | 1/51 (1) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-barr virus antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte morphology abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 3 (4) | 1 (1) | 4 (4) | 3 (4) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incoherent (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/85 (0) | 0/63 (0) | 1/51 (1) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/71 (0) | 0/38 (0) | 0/56 (0) | 0/43 (0) | 0/54 (0) | 0/239 (0) | 0/372 (0) | 0/248 (0) | 1/73 (1) | 0/105 (0) | 0/51 (0) | 0/8 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 1/404 (1) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 1/279 (1) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Vulva cyst (Reproductive system and breast disorders) | 0/85 (0) | 0/63 (0) | 0/51 (0) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 1/108 (1) | 0/43 (0) | 0/9 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 6 (6) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bereavement (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0/85 (0) | 0/63 (0) | 1/51 (1) | 0/58 (0) | 0/58 (0) | 0/279 (0) | 0/404 (0) | 0/265 (0) | 0/68 (0) | 0/108 (0) | 0/43 (0) | 0/9 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dialysis hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (6):
  • Study Protocol: Protocol J2W-MC-PYAB (m) (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/Prot_000.pdf
  • Study Protocol: PYAB 05 Protocol Addenda (2.2) (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/Prot_002.pdf
  • Study Protocol: J2W-MC-PYAB Addendum (4.2) (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/Prot_003.pdf
  • Statistical Analysis Plan: J2W-MC-PYAB Statistical Analysis Plan (V8) (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/SAP_001.pdf
  • Statistical Analysis Plan: J2W-MC-PYAB Statistical Analysis Plan Version 9 (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/SAP_004.pdf
  • Statistical Analysis Plan: J2W-MC-PYAB Statistical Analysis Plan A ddendum 4 (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04427501/SAP_005.pdf